CLINICAL TRIAL: NCT04446871
Title: Early Use of Methylene Blue in Patients With Septic Shock: a Pilot Randomized Controlled Trial
Brief Title: Methylene Blue in Early Septic Shock
Acronym: SHOCKEM-Blue
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Miguel Á Ibarra-Estrada, Principal investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCG/CEI-0252/17
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Septic Shock
Keywords: Septic shock; Methylene blue; Norepinephrine
MeSH Terms: conditions — Shock, Septic | interventions — Sodium Chloride; Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Placebo Comparator): Placebo
  Interventions: Drug: 0.9% sodium chloride
- Methylene blue (Experimental): Methylene blue
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: 0.9% sodium chloride — Intravenous infusion of 500 cc of 0.9% sodium chloride solution for 6 h, once a day for a total of 3 doses.
  Arms: Standard care
Drug: Methylene Blue — Intravenous infusion of 100 mg methylene blue in 500 cc of 0.9% sodium chloride solution for 6 h, once a day for a total of 3 doses.
  Arms: Methylene blue

SUMMARY:
Septic shock is a subset of sepsis characterized by a decrease in vascular tone, which contributes to impaired regional blood flow distribution, and leads to organic failure. Besides intravenous fluids and adequate antimicrobial therapy, patients with septic shock require vasopressor support, which can lead to many adverse effects, therefore, non-vasopressor agents that can improve hemodynamic status are needed. In this randomized controlled-study, the investigators will address the efficacy and safety of infusion with methylene blue in patients with septic shock.

DETAILED DESCRIPTION:
Unlike sepsis, septic shock mortality is not declining for the last decade, and is still around 40%. After restoring intravascular volume, many patients need vasopressor agents to maintain arterial blood pressure, which leads to improvement of perfusion at some vascular beds, however some organs may suffer from maldistribution of blood flow. These changes of regional blood flow may compromise oxygen delivery and perpetuate the inflammation and tissue damage associated with the state of shock.

One of the main mechanisms of vasodilation after inflammatory insults, is the activation of the inducible isoform of Nitric Oxide Synthase (iNOS), and the subsequent increase in the levels of nitric oxide, which even reduces the response to vasoconstrictor agents. Methylene blue (MB) is a selective inhibitor of iNOS, which has been used successfully in patients with post-cardiopulmonary bypass associated vasoplegia, however, the evidence of the use of MB in septic shock patients is limited to case reports, observational and small studies. In this randomized controlled trial, the investigators will compare the efficacy and safety outcomes of repeated doses of MB in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock diagnosis, according to the Sepsis-3 consensus.
* Prior adequate fluid resuscitation according to dynamic predictors of volume responsiveness.
* More than 6 h and less than 24 h of norepinephrine requirement to maintain a mean arterial pressure ≥65 mmHg.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Not expected to survive 48 hours.
* Presence or high suspicion of concurrent hemorrhagic, obstructive or hypovolemic shock.
* Personal or familiar history of glucose-6-phosphate dehydrogenase deficiency.
* Allergic to methylene blue, phenothiazines, or food dyes.
* Recent intake (4-weeks) of selective serotonin re-uptake inhibitors.
* Refusal of the patient or decision maker to enroll in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Vasopressor requirement | 28 days
  Total time to shock resolution (hours)

SECONDARY OUTCOMES:
Time to lactate normalization | 7 days
  Time in hours until lactate is <2 mmol/L
Length of stay in intensive care unit | 28 days
  Time in days until ICU discharge
Intensive care unit mortality | 28 days
  Mortality in intensive care unit

OTHER OUTCOMES:
Change in pulmonary function after treatment | 7 days
  Change in P/F index after three doses of methylene blue

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ibarra-Estrada, MD, Principal Investigator — Investigator
Locations (1):
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibarra-Estrada M, Kattan E, Aguilera-Gonzalez P, Sandoval-Plascencia L, Rico-Jauregui U, Gomez-Partida CA, Ortiz-Macias IX, Lopez-Pulgarin JA, Chavez-Pena Q, Mijangos-Mendez JC, Aguirre-Avalos G, Hernandez G. Early adjunctive methylene blue in patients with septic shock: a randomized controlled trial. Crit Care. 2023 Mar 13;27(1):110. doi: 10.1186/s13054-023-04397-7. PMID 36915146